CLINICAL TRIAL: NCT00147537
Title: A Phase 1b Dose Escalation/Phase 2 Randomized, Non-Comparative, Multiple Center, Open Label Study Of CP 751,871 In Combination With Paclitaxel And Carboplatin And Of Paclitaxel And Carboplatin Alone As First Line Treatment For Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Study Of CP-751,871 With Paclitaxel And Carboplatin In Advanced Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021002
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: non-small cell lung cancer; chemotherapy; figitumumab; insulin-like growth 1 factor receptor; IGF-IR; monoclonal antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — figitumumab; Paclitaxel; Carboplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 2 (Arms A & B) (Experimental): CP-751,871 + paclitaxel + carboplatin
  Interventions: Drug: CP-751,871; Drug: paclitaxel; Drug: carboplatin
- Phase 1b (Experimental): 1. Phase 1b Dose Escalation /Expansion: CP-751,871 + paclitaxel + carboplatin
  2. Phase 1b Erlotinib Extension: CP-751,871 + paclitaxel + carboplatin + erlotinib
  Interventions: Drug: CP-751,871; Drug: paclitaxel; Drug: carboplatin; Drug: erlotinib

INTERVENTIONS:
Drug: CP-751,871 — Phase 2 Arm A:
  CP-751,871 20 mg/kg IV over 2.5 hours up to 17 cycles
  Arms: Phase 2 (Arms A & B)
Drug: paclitaxel — Phase 2 Arm A:
  Paclitaxel 200 mg/m2, IV over 3 hours up to 6 cycles
  Phase 2 Arm B:
  Paclitaxel 200 mg/m2, IV over 3 hours up to 6 cycles
  Arms: Phase 2 (Arms A & B)
Drug: carboplatin — Phase 2 Arm A:
  Carboplatin AUC 6, IV over 15-60 minutes up to 6 cycles
  Phase 2 Arm B:
  Carboplatin AUC 6, IV over 15-60 minutes up to 6 cycles
  Arms: Phase 2 (Arms A & B)
Drug: CP-751,871 — Phase 1b Dose Escalation/Expansion: CP-751,871 20 mg/kg IV over 2.5 hours (up to 17 cycles) Phase 1b Erlotinib Extension: CP-751,871 20 mg/kg IV over 2.5 hours (up to 17 cycles)
  Arms: Phase 1b
Drug: paclitaxel — Phase 1b Dose Escalation/Expansion: paclitaxel 200 mg/m2, IV over 3 hours (up to 6 cycles) Phase 1b Erlotinib Extension: paclitaxel 200 mg/m2, IV over 3 hours (up to 6 cycles)
  Arms: Phase 1b
Drug: carboplatin — Phase 1b Dose Escalation/Expansion: carboplatin AUC 6, IV over 15-60 minutes (up to 6 cycles) Phase 1b Erlotinib Extension: carboplatin AUC 6, IV over 15-60 minutes (up to 6 cycles)
  Arms: Phase 1b
Drug: erlotinib — Phase 1b Erlotinib Extension: erlotinib 150 mg/day orally every day (up to 17 cycles)
  Arms: Phase 1b

SUMMARY:
Phase 1b Dose Excalation/Expansion: Identify and characterize safety and tolerability of recommended phase 2 dose of CP-751,871 when administered with paclitaxel and carboplatin Phase 1b Erlotinib Extension: To characterize the safety and tolerability of CP751,871 when administered with paclitaxel, carboplatin and erlotinib.

Phase 2: To test the efficacy of CP-751,871 combined with paclitaxel and carboplatin in the treatment of advanced non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/metastatic lung cancer

Exclusion Criteria:

* Previous treatment with chemotherapy
* Uncontrolled diabetes
* History/active cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2005-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (18):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shelbyville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Houston, Texas
- Pfizer Investigational Site, Montreal, Quebec, Canada
- Pfizer Investigational Site, Orbassano (TO), Italy
- Spain (3):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021002&StudyName=Combination%20Study%20Of%20CP-751%2C871%20With%20Paclitaxel%20And%20Carboplatin%20In%20Advanced%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 0.05 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 0.1 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 0.8 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 1.5 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 3 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 6 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 10 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 20 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b): Single intravenous (IV) dose of CP-751,871 20 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 1 year). Erlotinib 150 mg/day orally on Cycle 1 Day 1 (up to 1 year). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871(F)+Paclitaxel(P)+Carboplatin(C) (Phase 2): Single intravenous (IV) dose of CP-751,871 (F) 10 or 20 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each Cycle (up to 17 cycles). Paclitaxel (P) 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin (C) at dose to attain target area under the concentration-time curve (AUC) of 6 mg/mL*min, IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- Paclitaxel(P)+Carboplatin(C) (Phase 2): Paclitaxel (P) 200 mg/square meter (m^2) IV over 3 hours on Day 1 only of each cycle (up to 6 cycles) followed by carboplatin (C) at dose to attain target AUC of 6 mg/mL*min, IV over 15-60 minutes on Day 1 only of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
Period: Phase 1b
Arm/Group | CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b) | CP-751,871(F)+Paclitaxel(P)+Carboplatin(C) (Phase 2) | Paclitaxel(P)+Carboplatin(C) (Phase 2)
Started | 3 | 2 | 4 | 3 | 3 | 3 | 18 (18 participants randomized; 17 participants treated) | 7 | 18 (18 participants randomized; 17 participants treated) | 0 | 0
Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 2 | 2 | 4 | 2 | 3 | 3 | 18 | 7 | 17 | 0 | 0
Not completed — Death | 0 | 1 | 2 | 1 | 2 | 2 | 1 | 3 | 9 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 1 | 1 | 1 | 14 | 4 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Period: Phase 2
Arm/Group | CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b) | CP-751,871(F)+Paclitaxel(P)+Carboplatin(C) (Phase 2) | Paclitaxel(P)+Carboplatin(C) (Phase 2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 166 (166 particpants randomized; 163 participants treated) | 55 (55 randomized; 56 treated-1 randomized but not treated, 2 randomized to F+P+C rec'd P+C)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 161 | 52
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 85 | 31
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 47 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 4
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- CP-751,871 + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 0.05/0.1/0.8/1.5/3/6/10/20 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 + Paclitaxel + Carboplatin (Phase 2): Single intravenous (IV) dose of CP-751,871 10 or 20 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each Cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at dose to attain target area under the concentration-time curve (AUC) of 6 mg/mL*min, IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- Paclitaxel + Carboplatin (Phase 2): Paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 only of each cycle (up to 6 cycles) followed by carboplatin at dose to attain target AUC of 6 mg/mL*min, IV over 15-60 minutes on Day 1 only of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- Total: Total of all reporting groups
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2) | Total
Number analyzed (Participants) | 43 | 18 | 166 | 55 | 282
Age, Customized [Number; unit: participants]
  Less than 65 years old (<65) | 27 | 13 | 82 | 33 | 155
  65 to 69 years old (65 - 69) | 6 | 2 | 42 | 11 | 61
  70 years old and more than 70 years old (>=70) | 10 | 2 | 42 | 11 | 65
  Unspecified | 0 | 1 | 0 | 0 | 1
Sex/Gender, Customized [Number; unit: participants]
  Female | 18 | 8 | 49 | 21 | 96
  Male | 25 | 9 | 117 | 34 | 185
  Unspecified | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)of CP-751,871 in Combination With Paclitaxel and Carboplatin: Phase 1b
Description: The maximum tolerated dose of CP-751,871 in combination with paclitaxel and carboplatin is the highest dose level below the Maximum Administered Dose (the dose level at which 2 or more out of 3 to 6 patients experience a Dose Limiting Toxicity at a dose level in Cycle 1) at which none or one out of 6 patients experience a Cycle 1 Dose Limiting Toxicity.
Time Frame: Start of treatment (baseline) up to the end of Cycle 1 (Day 21)
Population: All participants who received at least one dose of any agent.
Measure: Number; unit: mg/kg
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 1b)
Number analyzed (Participants) | 42
mg/kg | NA — CP-751,871 was safe and well tolerated at dose levels up to 20 mg/kg, and MTD was not reached.

2. Primary Outcome: Recommended Phase 2 Dose (RP2D): Phase 1b
Time Frame: Start of treatment (baseline) up to the end of Cycle 1 (Day 21)
Population: All participants who received at least one dose of any agent.
Measure: Number; unit: mg/kg
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 1b)
Number analyzed (Participants) | 42
mg/kg | 20

3. Primary Outcome: Objective Response Rate: Phase 2
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: Every 2 cycles (7 to 10 days prior to the planned start of the next cycle, each cycle was 21 days) from start of treatment until either death or a total of 2 years from the date of randomization
Population: All participants who received any of the study treatments. N=number of participants who had measurable disease at baseline and an adequate baseline tumor assessment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 99 | 51
percentage of participants | 37.4 [29.2 to 46.1] | 27.5 [17.4 to 39.5]
Statistical Analysis 1: Comparison: CP-751,871 + Paclitaxel + Carboplatin (Phase 2); A one-sided p-value for H0: objective response rate <=0.28 using exact binomial test at level 0.05; Test type: Superiority or Other; p = 0.027, binomial test

4. Primary Outcome: Objective Response Rate in Non-Adenocarcinoma Participants: Phase 2
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2): Single intravenous (IV) dose of CP-751,871 20 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each Cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at dose to attain target area under the concentration-time curve (AUC) of 6 mg/mL*min, IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
Arm/Group | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 73
percentage of participants | 37.0 [27.5 to 47.2]
Statistical Analysis 1: Comparison: CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2); A One-sided p-value for H0: objective response rate <=0.30 using exact binomial test at level 0.05; Test type: Superiority or Other; p = 0.121, binomial test

5. Secondary Outcome: Objective Response Rate: Phase 1b
Description: as for outcome 3
Time Frame: as for outcome 3
Population: All participants who received at least one dose of any agent. N=number of participants who had measurable disease at baseline and an adequate baseline tumor assessment
Measure: Number; unit: percentage of participants
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 36 | 16
percentage of participants | 33.3 | 25.0

6. Secondary Outcome: Number of Participants With Positive Human Anti-human Antibody (HAHA) Values: Phase 1b
Description: HAHA are indicators of immunogenicity to CP-751,871.
Time Frame: Day 1 pre-infusion of each cycle up to Cycle 17 (each cycle was 21 day), 150 days after the last CP-751,871 infusion, and last follow up visit (one year post last study dose)
Population: All participants who received at least one dose of any agent. N=number of participants who were analyzed for HAHA
Measure: Number; unit: number of participants
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 21 | 8
number of participants | 1 | 0

7. Secondary Outcome: Number of Circulating Endothelial Cells (CECs): Phase 1b
Time Frame: Day 1 pre-dose and Days 15 to 21 of Cycle 4
Population: Per protocol amendment 6, blood samples for the rapid quantification of CECs were no longer collected from participants enrolled in the study. Insufficient data were available to evaluate for correlation.
Arm/Group | CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Circulating Tumor-Related Cells (CTCs) and CTC Insulin-Like Growth Factor 1 Receptor (IGF-IR) Expression: Phase 1b
Description: Blood samples were collected to enumerate the number of total CTCs and CTC insulin-like growth factor 1 receptor (IGF-IR) expression
Time Frame: Day 1 pre-dose and Days 15 to 21 of Cycle 4
Population: Per protocol amendment 6, blood samples for the rapid quantification of CTCs were no longer collected from participants enrolled in the study. Insufficient data were available to evaluate for correlation.
Arm/Group | CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Plasma Concentration of CP-751,871 at the End of Infusion (Cendinf) for Cycle 1 in Phase 1b
Time Frame: Cycle 1 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 2 pre-infusion (which is the end of Cycle 1)
Population: All participants who received at least one dose of each agent. N=number of participants contributing to the summary statistics
Measure: Mean (Standard Deviation); unit: milligram/liter (mg/L)
Groups:
- CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 0.8 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of Cycle 1 (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 1.5 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of Cycle 1 (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 6 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of Cycle 1 (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 10 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of Cycle 1 (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter*minute (mg/mL*min), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 4 | 3 | 3 | 3 | 14 | 6 | 16
milligram/liter (mg/L) | 1.510 | 17.34 (10.28) | 37.47 (9.0429) | 75.17 (22.250) | 147.3 (27.006) | 261.3 (62.278) | 415.7 (102.14) | 485.0 (131.83)

10. Secondary Outcome: Plasma Concentration of CP-751,871 at the End of Infusion (Cendinf) for Cycle 4 in Phase 1b
Time Frame: Cycle 4 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 8 | 3 | 9
mg/L | 2.975 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 19.15 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 40.70 | 100.7 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 327.0 | 331.1 (125.77) | 440.3 (211.67) | 447.3 (210.19)

11. Secondary Outcome: Area Under the Curve From Time Zero to 504 Hours [AUC (0-504)] Post Infusion of CP-751,871 for Cycle 1 in Phase 1b
Description: AUC (0-504)= Area under the plasma concentration versus time curve from time zero (pre-dose) to the end of the 21-day cycle, 504 hours(0-504)
Time Frame: Cycle 1 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 2 pre-infusion (which is the end of Cycle 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milligram.hour/Liter (mg.hr/L)
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 4 | 1 | 2 | 2 | 10 | 5 | 17
milligram.hour/Liter (mg.hr/L) | 22.30 | 2011 (1048.6) | 5320 | 12810 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 30500 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 54650 (14075) | 79820 (21767) | 85240 (33973)

12. Secondary Outcome: Area Under the Curve From Time Zero to 504 Hours [AUC (0-504)] Post Infusion of CP-751,871 for Cycle 4 in Phase 1b
Description: as for outcome 11
Time Frame: Cycle 4 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg.hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 2 | 0 | 2 | 1 | 7 | 1 | 6
mg.hr/L | 77.60 | 2410 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. |  | 23200 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 52500 | 94360 (11479) | 214000 | 133200 (21292)

13. Secondary Outcome: Area Under the Curve From Time Zero Extrapolated to Infinite Time [AUCinf] for CP-751,871 for Cycle 1 in Phase 1b
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) extrapolated to infinite time.
Time Frame: Cycle 1 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 2 pre-infusion (which is the end of Cycle 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg.hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 0 | 3 | 0 | 2 | 1 | 4 | 1 | 7
mg.hr/L |  | 1434 (914.58) |  | 16750 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 41200 | 69180 (10651) | 12100 | 107400 (37604)

14. Secondary Outcome: Plasma Decay Half-Life (t1/2) of CP-751,871 for Cycle 1 in Phase 1b
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Cycle 1 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 2 pre-infusion (which is the end of Cycle 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 0 | 3 | 0 | 2 | 1 | 4 | 1 | 7
Day |  | 2.84 (1.82) |  | 10.81 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 8.350 | 9.56 (2.02) | 11.10 | 9.89 (1.81)

15. Secondary Outcome: Plasma Decay Half-Life (t1/2) of CP-751,871 for Cycle 4 in Phase 1b
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Cycle 4 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4)
Population: as for outcome 9
Measure: Median (Standard Deviation); unit: Day
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Day |  | 5.360 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. |  |  | 15.40 |  |  |

16. Secondary Outcome: CP-751,871 Concentration at 504 Hours Post Dose (C504) for Cycle 1 (End of the 21-day Cycle) in Phase 1b
Description: Concentration at 504 hours post dose
Time Frame: Cycle 2 pre-infusion (which is the end of Cycle 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 0 | 4 | 1 | 2 | 2 | 11 | 5 | 17
mg/L |  | 0.1610 (0.3220) | 4.550 | 9.820 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 28.20 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 61.11 (23.125) | 95.20 (23.354) | 86.73 (57.117)

17. Secondary Outcome: CP-751,871 Concentration at 504 Hours Post Dose(C504) for Cycle 4 (End of the 21-day Cycle) in Phase 1b
Description: Concentration at 504 hours post dose
Time Frame: Cycle 5 pre-infusion (which is the end of Cycle 4)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 2 | 0 | 2 | 1 | 7 | 1 | 7
mg/L | 0.0000 | 0.4630 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. |  | 27.70 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 21.20 | 125.3 (16.101) | 357.0 | 158.6 (27.067)

18. Secondary Outcome: Accumulation of CP-751,871 Ratio (Cycle 4 AUC504 / Cycle 1 AUC504) (Rac) in Phase 1b
Description: Accumulation ratio (Cycle 4 AUC504 / Cycle 1 AUC504) (Rac)
Time Frame: Cycle 1 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 2 pre-infusion (which is the end of Cycle 1). Cycle 4 pre-infusion, 1 and 24 hour and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4).
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 2 | 0 | 2 | 1 | 7 | 1 | 6
ratio | 3.480 | 1.009 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. |  | 1.830 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 1.550 | 1.984 (0.3015) | 2.260 | 1.962 (0.4283)

19. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration of CP-751,871(AUClast) for Cycle 1 in Phase 1b
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Cycle 1 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 2 pre-infusion (which is the end of Cycle 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg.hr/L
Groups:
- CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b): Single intravenous (IV) dose of CP-751,871 0.05 milligram/kilogram (mg/kg) over 2.5 hours on Day 1 of each cycle (up to 17 cycles). Paclitaxel 200 mg/square meter (m^2), IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 6 milligram/milliliter (mg/mL), IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 4 | 3 | 3 | 3 | 12 | 6 | 17
mg.hr/L | 16.60 | 1235 (713.55) | 5137 (1682.5) | 11350 (5551.7) | 25630 (12536) | 49260 (18770) | 71200 (26855) | 87680 (35247)

20. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration of CP-751,871 (AUClast) for Cycle 4 in Phase 1b
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Cycle 4 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg.hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 2 | 1 | 2 | 1 | 9 | 3 | 9
mg.hr/L | 64.70 | 2255 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 2670 | 23400 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 70300 | 82930 (29539) | 116200 (83683) | 114000 (44197)

21. Secondary Outcome: Maximum Observed Plasma CP-751,871 Concentration (Cmax) for Cycle 1 in Phase 1b
Description: Maximum Observed Plasma Concentration
Time Frame: Cycle 1 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 2 pre-infusion (which is the end of Cycle 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 1 | 4 | 3 | 3 | 3 | 14 | 6 | 17
mg/L | 1.510 | 17.34 (10.280) | 38.60 (10.989) | 75.17 (22.250) | 147.3 (27.006) | 275.2 (89.932) | 415.7 (102.14) | 483.1 (128.14)

22. Secondary Outcome: Maximum Observed Plasma CP-751,871 Concentration (Cmax) for Cycle 4 in Phase 1b
Description: Maximum Observed Plasma Concentration
Time Frame: Cycle 4 pre-infusion, 1 and 24 hours and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is then end of Cycle 4)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b)
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 9 | 3 | 10
mg/L | 2.975 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 20.25 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 40.70 | 100.7 (NA) — As planned, standard deviation was not calculated for the groups with fewer than 3 participants analyzed. | 327.0 | 369.1 (91.602) | 611.3 (43.501) | 535.5 (180.97)

23. Secondary Outcome: Number of Participants With Positive Human Anti-human Antibody (HAHA) Values: Phase 2
Description: HAHA are indicators of immunogenicity to CP-751,871
Time Frame: Day 1 pre-infusion of each Cycle (each cycle was 21 day) up to Cycle 17 and 150 days after the last CP-751,871 infusion
Population: All participants who received any of the study treatments. N=number of participants who were analyzed for HAHA
Measure: Number; unit: number of participants
Groups:
- Paclitaxel + Carboplatin + Additional CP-751,871 (Phase 2): Paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 only of each cycle (up to 6 cycles) followed by carboplatin at dose to attain target AUC of 6 mg/mL, IV over 15-60 minutes on Day 1 only of each cycle (up to 6 cycles). Each cycle was 21 day cycle. Participants that were considered to be in stable disease after at least 4 cycles of treatment or in progressive disease at any time during the study could receive additional cycles of treatment with CP-751,871 in combination with Paclitaxel and Carboplatin or CP-751,871 alone.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin + Additional CP-751,871 (Phase 2)
Number analyzed (Participants) | 38 | 4
number of participants | 0 | 0

24. Secondary Outcome: M.D. Anderson Symptom Assessment Inventory (MDASI) in Phase 2
Description: The MDASI is a 19-item questionnaire that assesses the severity of 13 symptoms over the past 24 hours, as well as how much the symptoms interfered with 6 areas of function (eg, walking, work, mood), when the symptom was "at its worst". Each item is scored from 0 to 10, with '0' indicating that the symptom was either not present or did not interfere with their activities, and '10' indicating that the symptom was "as bad as you can imagine" or "interfered completely" with their life. Total average score range: 0 to 10.
Time Frame: Day 1 pre-dose of Cycle 1, weekly for Cycle 1 and 2, monthly prior to each subsequent cycle (Cycle 3 up to Cycle 17, each cycle was 21 day), and follow up (one year post last study dose)
Population: Due to the status of the program, no participants were analyzed for MDASI in phase 2.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Version 3.0 (EORTC-QLQ-C30/-LC13) in Phase 2
Description: The QLQ-C30/-LC13 is a 43 item, self-administered questionnaire designed to assess health outcomes in clinical trials. In addition to global quality of life, the measure assesses 5 functional domains (physical, role, cognitive, emotional and social functioning) and specific symptoms (eg, nausea, pain). Each item is rated on a 1-4 scale with '1' representing "not at all" and '4' "very much". Within domains, items are scored to obtain a total score with higher scores representative of poorer HRQoL. Scale score range: 0 to 100.
Time Frame: Day 1 pre-dose of Cycle 1, monthly prior to each cycle (up to 17 cycles, each cycle was 21 day), and follow up (one year post last study dose)
Population: Due to the status of the program, no participants were analyzed for EORTC-QLQ-C30/-LC13 in phase 2.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Apparent Volume of CP-751,871 Distribution (Vd) for Cycle 4 in Phase 2
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Cycle 4 pre-infusion, 1 and 24 hour and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4)
Population: Volume of distribution (Vd) was not calculated based on the status of the program and the limited value this further pharmacokinetic analyses would provide.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Clearance (CL) of CP-751,871 for Cycle 4 in Phase 2
Description: Systemic clearance.
Time Frame: Cycle 4 pre-infusion, 1 and 24 hour and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4).
Population: Clearance (CL) were not calculated based on the status of the program and the limited value this further PK analyses would provide.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Area Under the Curve From Time Zero to 504 Hours [AUC (0-504)] Post Infusion of CP-751,871 for Cycle 4 in Phase 2
Description: as for outcome 11
Time Frame: Cycle 4 pre-infusion, 1 and 24 hour and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4).
Population: AUC504 was not calculated for Cycle 4 in Phase 2 based on the status of the program and the limited value this further PK analyses would provide.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: CP-751,871 Concentration at 504 Hours Post Dose(C504) for Cycle 4 (End of the 21-day Cycle) in Phase 2
Description: Concentration at 504 hours post dose
Time Frame: Cycle 4 pre-infusion, 1 and 24 hour and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4).
Population: C504 was not calculated for Cycle 4 in Phase 2 based on the status of the program and the limited value this further PK analyses would provide.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Maximum Observed Plasma CP-751,871 Concentration (Cmax) for Cycle 4 in Phase 2
Description: Maximum Observed Plasma Concentration
Time Frame: Cycle 4 pre-infusion, 1 and 24 hour and 4 and 8 days post infusion, Cycle 5 pre-infusion (which is the end of Cycle 4).
Population: Cmax was not calculated for Cycle 4 in Phase 2 based on the status of the program and the limited value this further PK analyses would provide.
Arm/Group | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2)
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Progression-Free Survival (PFS): Phase 2
Description: Time in months from start of study treatment to first documentation of objective tumor progression or death due to any cause whichever comes first. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression was determined from radiological image (where data meet the criteria for progressive disease [PD]).
Time Frame: as for outcome 3
Population: All participants who received any of the study treatments.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 2): Single intravenous (IV) dose of CP-751,871 10 mg/kg IV over 2.5 hours on Day 1 of each Cycle (up to 17 cycles). Paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at dose to attain target AUC of 6 mg/mL*min, IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
- CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2 NR): Phase 2 Non-Randomized (NR) Extension Cohort. Single intravenous (IV) dose of CP-751,871 20 mg/kg IV over 2.5 hours on Day 1 of each Cycle (up to 17 cycles). Paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 of each cycle (up to 6 cycles) followed by carboplatin at dose to attain target AUC of 6 mg/mL*min, IV over 15-60 minutes on Day 1 of each cycle (up to 6 cycles). Each cycle was 21 days cycle.
Arm/Group | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 2) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2 NR)
Number analyzed (Participants) | 58 | 49 | 56 | 56
months | 4.4 [3.8 to 5.6] | 4.5 [3.9 to 5.6] | 4.3 [3.9 to 5.4] | 5.1 [4.0 to 5.8]

32. Secondary Outcome: Time to Progression (TTP) in Phase 2
Description: Time in months from start of study treatment to first documentation of objective tumor progression. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression was determined from radiological image (where data meet the criteria for progressive disease [PD]).
Time Frame: as for outcome 3
Population: Due to the status of the program, time to progression was not was not analyzed.
Arm/Group | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 2) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2 NR)
Number analyzed (Participants) | 0 | 0 | 0 | 0

33. Secondary Outcome: Duration of Response (DR) in Phase 2
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.44. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 3
Population: Due to the status of the program, duration of response was not analyzed.
Arm/Group | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 2) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 2 NR)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b) | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin (Phase 2) | Paclitaxel + Carboplatin + Additional CP-751,871 (Phase 2)
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2 | 2/4 | 1/3 | 2/3 | 2/3 | 7/17 | 2/7 | 9/17 | 86/163 | 9/56 | 3/22
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 4/4 | 3/3 | 3/3 | 3/3 | 17/17 | 7/7 | 17/17 | 162/163 | 55/56 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=2) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=4) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=17) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=7) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b) (N=17) | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) (N=163) | Paclitaxel + Carboplatin (Phase 2) (N=56) | Paclitaxel + Carboplatin + Additional CP-751,871 (Phase 2) (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 11 | 2 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 12 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 11 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic complication (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catatonia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Personality disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 0.05 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 0.1 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=2) | CP-751,871 0.8 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=4) | CP-751,871 1.5 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 3 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 6 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=3) | CP-751,871 10 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=17) | CP-751,871 20 mg/kg + Paclitaxel + Carboplatin (Phase 1b) (N=7) | CP-751,871 + Paclitaxel + Carboplatin + Erlotinib (Phase 1b) (N=17) | CP-751,871 + Paclitaxel + Carboplatin (Phase 2) (N=163) | Paclitaxel + Carboplatin (Phase 2) (N=56) | Paclitaxel + Carboplatin + Additional CP-751,871 (Phase 2) (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 4 | 9 | 56 | 15 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 13 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 6 | 0 | 6 | 52 | 13 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 43 | 12 | 3
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 8 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 17 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 2 | 49 | 17 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 2 | 2 | 9 | 3 | 11 | 65 | 12 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 11 | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 4 | 1 | 0 | 19 | 5 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 15 | 1 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 7 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3 | 0 | 10 | 2 | 11 | 84 | 24 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 4 | 1 | 7 | 30 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 5 | 2 | 9 | 48 | 11 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 6 | 27 | 5 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 18 | 1 | 2
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 1
Fatigue (General disorders) | 3 | 2 | 1 | 3 | 3 | 2 | 10 | 5 | 8 | 107 | 26 | 14
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 8 | 27 | 5 | 2
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 6 | 5
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 17 | 7 | 2
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 24 | 7 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 2 | 3
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 8 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pneumonia 1 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 2 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 5
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 8 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 16 | 2 | 2
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 10 | 2 | 1
Blood alkaline phosphatase (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 0
Blood creatinine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Blood lactate dehydrogenase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 11 | 6 | 5
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 0 | 2
Gamma-glutamyltransferase (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 27 | 6 | 2
Haemoglobin (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 10 | 4 | 4
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 5 | 4 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 5 | 9 | 4 | 3
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Troponin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 5 | 1 | 6 | 35 | 2 | 4
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4 | 3 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 9 | 2 | 8 | 69 | 15 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 14 | 2 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 6 | 3 | 11 | 67 | 9 | 8
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 10 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 6 | 4 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 17 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 0 | 2 | 6 | 3 | 8 | 48 | 18 | 7
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 25 | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 7 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 4 | 15 | 3 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 7 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 18 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 7 | 32 | 13 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 4 | 0 | 1 | 27 | 6 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 4 | 27 | 4 | 4
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 5 | 4 | 5 | 43 | 7 | 6
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 30 | 2 | 4
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 6 | 3 | 4 | 57 | 22 | 14
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 16 | 4 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 5 | 38 | 10 | 2
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 9 | 4 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 7 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 5 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 13 | 4 | 3
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 9 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scrotal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 4 | 2 | 3 | 35 | 7 | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 3 | 5 | 40 | 15 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 5 | 26 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 20 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 4 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 5 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 2 | 3 | 3 | 10 | 3 | 10 | 91 | 31 | 15
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 2 | 7 | 10 | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 9 | 0 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 8 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 5 | 1 | 13 | 33 | 4 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 5 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 11 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental plaque (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gravitational oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 2
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear lobe infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 1 | 1
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 1 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Blood immunoglobulin G increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coagulation test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematocrit (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio normal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Red blood cell sedimentation rate (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin I (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urinary casts (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urine leukocyte esterase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Hyperphagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonic convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vocal cord paralysis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Denture wearer (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.